CLINICAL TRIAL: NCT06810232
Title: Effects of General Health Risk Factors on Prolonged Hospital Stay in Non-operating Room Anesthesia Preoperative Anesthesia Examination; Prospective Study
Brief Title: Effects of General Health Risk Factors on Prolonged Hospital Stay
Status: Enrolling by invitation | Type: Observational
Sponsor: Naime Yalçın (Other)
Responsible Party: Sponsor-Investigator, Naime Yalçın, Specialist Anesthesiology and Reanimation, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2024.12.276
Record Dates: First submitted 2025-01-27; First posted 2025-02-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Preoperative Evaluation; Anesthesia; Day Surgery; Life Style; Hospital Stay
MeSH Terms: interventions — Endoscopy, Gastrointestinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General health risk factors: Arm HT, Arm DM, Arm Asthma, Arm Obezity, Arm Immobility, Arm Smoke
  Interventions: Procedure: Gastrointestinal endoscopy

INTERVENTIONS:
Procedure: Gastrointestinal endoscopy — Patients will be divided into groups according to general health risk factors detected during preoperative anesthesia evaluation (hypertension, diabetes, asthma, obesity, chronic disease, medication history, immobility, smoking, etc.) and will be evaluated in terms of age, gender, weight and height will be combined to report BMI in kg/m2, alcohol, allergy, ASA, endoscopy site, complications that may develop related to anesthesia and sedation (such as hemodynamic instability, hemoglobin desaturation, pulmonary aspiration and apnea), additional interventions, and hospital stay.

SUMMARY:
According to the literature, a detailed preoperative anesthesia assessment systematically verifies perioperative risks, provides functional and physiological optimization, improves the patient's condition and the perioperative process, and prevents complications. In this context, the investigators aimed to determine the frequency of lifestyle risk factors in patients who applied to investigator's clinic for preoperative anesthesia assessment due to adult gastrointestinal endoscopy, to investigate the relationship between lifestyle risk factors and factors and outcomes during the anesthesia procedure, and to compare the effects of these risk factors on developing complications and hospital stay.

DETAILED DESCRIPTION:
A detailed preoperative anesthesia assessment systematically validates perioperative risks, optimizes functional and physiological functions, improves patient status and perioperative process, and prevents complications. Preoperative anesthesia assessment clinics are an ideal environment to examine patients' medical conditions, ensure patient safety, and maximize economic efficiency in the preoperative period. The number of procedures performed in outpatient surgery centers has now far exceeded inpatient procedures. With an estimate that 44% of increasingly difficult adverse perioperative events are preventable, it is anticipated that perioperative complications can be reduced through anesthesia clinic examinations. In the absence of clinical examinations, surgical delays and case cancellations due to incomplete patient information will occur. In recent years, the implementation of a large number of complex surgical procedures and the planning of more complicated patients for intervention in the outpatient setting have contributed significantly to the development of day surgery. With the significant increase in the number of patients undergoing outpatient surgery, comprehensive and detailed preoperative assessment and optimization have become increasingly important in patients with multiple comorbidities and unusual conditions. Preoperative screening is essential for patients at risk who may benefit from preoperative optimization. For this purpose, close communication between the surgeon, anesthesiologist, and family physician is essential. There is no doubt that perioperative morbidity and mortality are closely related to the patient's preoperative health status, the surgical procedure performed, and the anesthesia technique used. Various studies have been conducted to confirm and quantify the relationships between risk factors and the incidence of perioperative adverse events. Perioperative factors, accompanied by preoperative risk assessment, help identify patients at increased risk and enable management strategies to reduce postoperative complications and improve patient outcomes. Anesthesia services for gastrointestinal (GI) endoscopic procedures are included in outpatient anesthesia procedures and have increased significantly in frequency over the years. Before 2004, only a fraction of endoscopic procedures were performed with anesthesia, while by 2009, 30-35% of upper endoscopy and colonoscopies were performed with anesthesia under sedation, and this number increased to half of colonoscopies in 2012. Although the use of propofol in endoscopic surgery has increased, the relationship between increased complications due to sedation remains unclear. While some studies have reported increased risk of aspiration pneumonia, colon perforation, bleeding, and cardiovascular events, other studies have shown that there is no increase in the risk of complications during this process. The primary aim of investigator's study was to determine the frequency of lifestyle risk factors in patients who applied to investigator's clinic for preoperative anesthesia evaluation due to adult gastrointestinal endoscopy. Secondarily, the investigator aimed to compare the effects of these risk factors on complications and hospital stay by investigating the relationship between lifestyle risk factors and factors and outcomes during the anesthesia procedure.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* ASA I-IV status
* Undergoing surgery for gastrointestinal endoscopy
* Under sedation anesthesia

Exclusion Criteria:

* In case the procedure is performed while awake
* Emergency endoscopy
* ASA-E is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who apply to our hospital's anesthesia outpatient clinic for preoperative anesthesia evaluation for gastrointestinal endoscopy.
Sampling Method: Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Association between general health risk factors and prolonged hospital stay | Up to 8 weeks after registration
  Investigator planned to divide patients who applied to investigator's anesthesia clinic for gastrointestinal endoscopy into groups according to their general health risk factors (hypertension, diabetes, asthma, immobility, obesity, smoking, etc.) during preoperative anesthesia evaluations, and to primarily determine the number of patients who admitted in the ward after endoscopy despite performing day-case procedures among the groups, and secondarily, to observe the frequency of endoscopy procedures for each group, as well as to examine the length of stay in the recovery unit and complications after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)